CLINICAL TRIAL: NCT01739439
Title: RT-054: A Phase I Study of Neoadjuvant Hypofractionated Chemoradiation Plus Radiosurgical Boost for Patients With Borderline Resectable and Locally Advanced Unresectable Pancreatic Cancer
Brief Title: Chemoradiation and Radiosurgery Boost in Treating Patients With Locally Advance Pancreatic Cancer That May or May Not be Removed by Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-046; NCI-2012-02729 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radiotherapy, Intensity-Modulated; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemoradiation and radiosurgery) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes once weekly and undergo hyperfractionated IMRT 5 days a week in weeks 1-3. Patients then undergo a single fraction of radiosurgery boost in week 5 and then receive gemcitabine hydrochloride IV over 30 minutes once weekly in weeks 6-8. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Radiation: hyperfractionated radiation therapy; Radiation: intensity-modulated radiation therapy; Radiation: radiosurgery; Procedure: diffusion-weighted magnetic resonance imaging

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Radiation: hyperfractionated radiation therapy — Undergo hyperfractionated IMRT
Radiation: intensity-modulated radiation therapy — Undergo hyperfractionated IMRT
  Other Names: IMRT
Radiation: radiosurgery — Undergo radiosurgery boost
  Other Names: radiation surgery
Procedure: diffusion-weighted magnetic resonance imaging — Correlative studies
  Other Names: diffusion-weighted MRI

SUMMARY:
This phase I trial studies the side effects and best dose of radiosurgery boost following chemoradiation in treating patients with locally advanced pancreatic cancer that may or may not be removed by surgery. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Radiosurgery can send x-rays directly to the tumor and cause less damage to normal tissue. Giving chemotherapy and radiation therapy together with radiosurgery may kill more tumor cells and allow doctors to save the part of the body where the cancer started

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of a radiosurgery boost added to hypofractionated chemoradiation in patients with borderline resectable or unresectable pancreatic cancer.

SECONDARY OBJECTIVES:

I. To determine the effect of a radiosurgery boost added to hypofractionated chemoradiation on surgical morbidity (specifically, healing of the surgical anastomoses and abdominal wounds and late hemorrhage from blood vessels in the field) in patients with advanced borderline resectable (BLR) or unresectable pancreatic cancer.

II. To evaluate the utility of diffusion-weighted magnetic resonance imaging (MRI) as an assessment of treatment response after chemoradiation followed by radiosurgery.

III. To determine the feasibility of collecting tissue for immunohistochemistry (IHC) analysis via endoscopic ultrasound or computed tomography (CT)-guided fine needle aspiration.

IV. To utilize pathologic response rates in dose escalated regions, hypofractionated regions, and the dose gradient region in between to better characterize the radiobiologic response of pancreatic cancer to radiation dose escalation.

OUTLINE: This is a dose-escalation study of radiosurgery.

Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes once weekly and undergo hyperfractionated intensity-modulated radiation therapy (IMRT) 5 days a week in weeks 1-3. Patients then undergo a single fraction of radiosurgery boost in week 5 and then receive gemcitabine hydrochloride IV over 30 minutes once weekly in weeks 6-8. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically-confirmed pancreatic adenocarcinoma
* For the initial dose escalation study, patients must have locally advanced / unresectable pancreatic cancer; these are defined as follows:

  * No distant metastases
  * Hepatic artery encasement
  * Superior mesenteric artery (SMA) encasement > 180 degrees
  * Any celiac axis abutment
  * Unreconstructable superior mesenteric vein (SMV)/portal occlusion
  * Aortic invasion or encasement
  * Metastases to lymph nodes beyond the field of resection
* For the expansion phase, patients must have borderline resectable or locally advanced / unresectable pancreatic cancer; these are defined as follows:

  * No distant metastases
  * At least 45 degree abutment of the hepatic artery or SMA
  * Any celiac axis abutment
  * Near complete occlusion of the SMV or portal vein
  * Unreconstructable or reconstructible SMV/portal occlusion
  * Aortic invasion or encasement
  * Metastases to lymph nodes beyond the field of resection
* Patients must have evaluable disease
* Women of childbearing potential must be non-pregnant (negative pregnancy test within 72 hours prior to radiation simulation, postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential) and nonlactating, and men and women must be willing to exercise an effective form of birth control (abstinence/contraception) while on study and for 3 months after therapy completed
* Eastern Cooperative Oncology Group (ECOG) performance status determined to be between 0 and 1
* Absolute neutrophil count (ANC) >= 1,500/ul
* Platelets (PLT) >= 100,000/ul
* Subjects must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up
* Bilirubin less then 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN
* Serum creatinine < 1.5 x ULN

Exclusion Criteria:

* Patients who have had any prior therapy for pancreatic cancer
* Concurrent chemotherapy or biologic therapy
* A history of ataxia telangiectasia or other documented history of radiation hypersensitivity
* Scleroderma or active connective tissue disease
* Active inflammatory bowel disease
* Serious, active infections requiring treatment with IV antibiotics
* Uncontrolled intercurrent illness including, but not limited to, psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level in which 1 out of 6 patients observes dose-limiting toxicity (DLT) assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meyer, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States